CLINICAL TRIAL: NCT04683120
Title: Real-time Diagnosis and Visualization of Tumor Margins in Excised Breast Specimens Using Zenith FLIM Diagnostics
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: New Medical Team and Surgical Center Location
Sponsor: Laser LabCorp (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Laser LabCorp #001
Record Dates: First submitted 2020-12-19; First posted 2020-12-24 (Actual); Last update posted 2021-06-30 (Actual); Status verified 2021-06

CONDITIONS: Oncology; Breast Cancer; Cancer Diagnosis; Margins of Excision; Margins, Tumor-Free
Keywords: Oncology; Breast Cancer; Zenith FLIM Diagnostics; FLIM; Tumor; Margin Assessment
MeSH Terms: conditions — Neoplasms; Breast Neoplasms; Margins of Excision

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Arm Study (Experimental): This is a single arm study, which will involve all patients qualifying for Breast Conservation Therapy as a part of their breast cancer management excluding patients undergoing neoadjuvant therapy for inoperable disease.
  Interventions: Diagnostic Test: Zenith FLIM Diagnostics

INTERVENTIONS:
Diagnostic Test: Zenith FLIM Diagnostics — In-vitro

SUMMARY:
Our investigational team has developed a technology to visualize the operative margins in 'real time,' in other words during the operation while the patient is still on the table. While different surgeons use different operative techniques, our technique involves removing the main lumpectomy specimen, marking two of its borders with suture to orient the specimen for correct pathologic evaluation.

The FLIM (Fluorescent Lifetime Imaging Microscopy) technique can differentiate between cancerous and noncancerous specimens using a complex algorithm that essentially utilizes a definitive delta between the metabolic activities of diseased and non-diseased tissue. The research coordinator along with the surgeon will be able to insert the lumpectomy specimen followed by the 6 shaved margins (one by one) in a matter of minutes once the specimens have been resected. To be clear, the FLIM analysis will be taking place in- vitro. The device is invitro test and would be tested against the gold standard the pathologist biopsy.

FLIM analysis by the surgeon will not take more than several minutes, therefore not adding any significant time for patient to be under anesthesia. All specimens will be removed from the patient's body prior to their evaluation by the FLIM technique. Our team will not be making decisions based on FLIM analysis during this early phase of study. In other words, even if FLIM suggests a positive margin still exists in the body, our team will not act on these results by resecting additional tissue at this stage. FLIM margin results will be compared directly with pathology results for accuracy of the findings.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the effectiveness of the investigational Zenith FLIM Diagnostics imaging device that's modality is a direct support during lumpectomy cancer surgery to achieve the common goal of improving patient quality of life by decreasing rates of re-operation. The team is fully dedicated to bringing the Gold Standard in the operating room, enabling margin assessment, in real time, at the histological detail.

Our operative technique involves removing the main lumpectomy specimen, marking two of its borders with suture to orient the specimen for correct pathologic evaluation. Next, we take 6 shave margins in all directions around the lumpectomy cavity (superior, inferior, medial, lateral, posterior, anterior) and anchor an orientation stitch at the far side of the margin, again, for pathologist to understand which side was farthest away from the lumpectomy specimen.

The research coordinator along with the surgeon will be able to insert the lumpectomy specimen into the Zenith FLIM device followed by the 6 shaved margins (one by one) in a matter of minutes once the specimens have been resected. To be clear, the Zenith FLIM analysis will be taking place in-vitro. The machine will be placed a good distance from the patient, in an ante-room, and does not require sterility. Of course, if the surgeon breaks sterility while handing off the specimens for FLIM analysis, he or she will have to re-sterilize as would be standard if sterile conditions are broken for any other reasons (having to re-scrub because sterility is broken is a common procedure). Once the specimens are placed in the Zenith FLIM, the specimens will no longer be sterile, but there is no need to maintain sterility of the specimens once they are in-vitro. In fact, even in the absence of Zenith FLIM analysis, once the specimens are placed in cups for pathologic evaluation, they are no longer sterile. In other words, loss of sterility of the specimen is a necessity of the operation regardless of Zenith FLIM analysis.

The device is an in-vitro test and would be tested against the gold standard: the pathologic evaluation of resected tissue. The test results would not be used for any diagnosis. Neither the test nor the unit comes in contact with patients under any circumstance. The Zenith FLIM margin results will be compared directly with pathology. The effectiveness of the Zenith FLIM Diagnostics margin results will be compared directly with pathology and evaluated in this study.

ELIGIBILITY:
Inclusion Criteria:

* A) Age18 and over
* B) EnglishSpeaking
* C) Able to read and understand consent
* D) All patient's candidate for lumpectomy
* E) Recurrent cancer patients requiring lumpectomy
* F) All stages and grades of cancer as long as patient is lumpectomy candidate
* G) Margin1(S)
* H) Margin 2(I)
* I) Margin 3 (M)
* J) Margin 4 (L)
* K) Margin5(P)
* L) Margin 6 (A)

Exclusion Criteria: Exclusion criteria includes any patients with autoimmune disease affecting breast tissue anyone receiving neoadjuvant chemotherapy prior to lumpectomy, any patient undergoing mastectomy.

* A) Extensively damaged tissue
* B) Abnormal tissue(auto immune disease)
* C) Neoadjuvant treated breast
* D) Mastectomy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-12-15 (Estimated); Primary Completion 2022-08-03 (Estimated); Study Completion 2022-11-02 (Estimated)

PRIMARY OUTCOMES:
Tumor Distance From Margins in all 6 Dimensions | 5-10 minutes after tumor and margins are extricated from body
  Tumor distance from margin in all 6 dimensions compared to final histopathologic diagnosis/confirmation in testing for accuracy of the Zenith FLIM.

CONTACTS AND LOCATIONS:
Overall Officials: Brad Schoengood, Study Chair — Laser LabCorp
Locations (1):
- Laser LabCorp, New York, New York, United States